CLINICAL TRIAL: NCT00774800
Title: Phase II Study Evaluating Pharmacokinetics and Postprandial Glycemic Response of Subcutaneously Injected Humalog and Humulin R With/Without Co-Injected Recombinant Human Hyaluronidase Following Liquid Meal in Type1 Diabetes Mellitus Patients
Brief Title: Phase II Pharmacokinetics Study of Humalog and Humulin-R With and Without rHuPH20 in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HZ2-08-05; HALO-117-201 (Other: Halozyme Therapeutics, Inc.)
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Recombinant Hyaluronidase; Type 1 Diabetes Mellitus; Humalog; Humulin R; rHuPH20; Hylenex
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Lispro; Insulin; Insulin, Regular, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- First Humalog+PH20, then Humalog, Humulin-R+PH20, Humulin-R (Experimental): Humalog + Recombinant human hyaluronidase PH20 (rHuPH20) (Intervention 1): 24 units (U) of rHuPH20 per unit of Humalog, injected subcutaneously (SC), for up to 3 visits until an appropriate dose was identified.
  Humalog alone (Intervention 2): a single SC injection of the appropriate identified dose of Humalog, delivered before a liquid meal.
  Humulin-R + rHuPH20 (Intervention 3): 24 U of rHuPH20 per unit of Humulin-R, injected SC, for up to 2 visits until an appropriate dose was identified.
  Humulin-R alone (Intervention 4): a single SC injection of the appropriate identified dose of Humulin-R, delivered before a liquid meal.
  Appropriate dose of either Humalog or Humulin-R was that at which blood glucose following a liquid meal was <160 milligrams per deciliter (mg/dL) for more than 30 minutes during the first 4 hours after injection and never fell below 60 mg/dL.
  All dose finding visits and interventions were separated by 3-10 days.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20); Other: Liquid meal

INTERVENTIONS:
Drug: Humalog
  Other Names: Insulin lispro
Drug: Humulin-R
  Other Names: Humulin; Recombinant human insulin
Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
  Other Names: HYLENEX; PH20
Other: Liquid meal
  Other Names: Ensure

SUMMARY:
Humalog and Humulin-R (recombinant human insulin) are Food and Drug Administration (FDA) approved medications for the treatment of diabetes mellitus. Recombinant human hyaluronidase PH20 (rHuPH20) is approved by the FDA for use as an aid in the absorption and dispersion of other injectable drugs. In this study, rHuPH20 will be co-administered with both Humalog and Humulin-R in order to determine if it improves the absorption of these insulins to more closely mimic the body's natural increase in insulin in response to a meal.

DETAILED DESCRIPTION:
Participants received all 4 interventions in the same order.

Dose-finding visits were conducted to identify the appropriate dose of Humalog and Humulin-R. For each Humalog dose-finding visit, a total of 24 U of rHuPH20 was injected SC per unit of Humalog, corresponding to a mass concentration of 18.2 micrograms per milliliter (μg/mL) rHuPH20 (at final concentration of 91 U/mL of Humalog). For each Humulin-R dose-finding visit, a total of 24 U of rHuPH20 was injected SC per unit of Humulin-R, corresponding to a mass concentration of 20.0 μg/mL rHuPH20 (at final concentration of 100 U/mL of Humulin-R).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age 18 to 65 years, inclusive. Females of child-bearing potential must use a standard and effective means of birth control for the duration of the study.
* Participants with Type 1 diabetes mellitus treated with insulin for greater than or equal to 12 months.
* Body mass index (BMI) 18.0 to 29.0 kilograms per meter squared (kg/m^2), inclusive.
* Glycosylated hemoglobin A1c (HbA1c) less than or equal to 10% based on local laboratory results.
* Fasting C-peptide less than 0.6 nanograms per milliliter (ng/mL).
* Current treatment with insulin less than 1.2 units per kilogram per day (U/kg/day).
* Participants should be in good general health based on medical history and physical examination, without medical conditions that might prevent the completion of study drug injections and assessments required in this protocol.

Exclusion Criteria:

* Known or suspected allergy to any component of any of the study drugs in this trial.
* Previous enrollment in this trial.
* A participant who has proliferative retinopathy or maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
* Clinically significant (as judged by the Investigator) active disease of the gastrointestinal, cardiovascular (including a history of arrhythmia or conduction delays on electrocardiogram [ECG]), hepatic, neurological, renal, genitourinary, or hematological systems, or uncontrolled hypertension (diastolic blood pressure greater than or equal to 100 millimeters of mercury [mmHg] and/or systolic blood pressure greater than or equal to 160 mmHg after 5 minutes in the supine position).
* History of any illness or disease that in the opinion of the Investigator might confound the results of the trial or pose additional risk in administering the study drugs to the participant.
* Clinically significant findings (as judged by the Investigator) in routine laboratory data, including anemia with hemoglobin less than lower limits of normal at screening.
* Use of drugs which may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia.
* Recurrent major hypoglycemia or hypoglycemic unawareness, as judged by the Investigator.
* Current addiction to alcohol or substances of abuse as determined by the Investigator.
* Blood donation (>500 milliliters [mL]) within the 9 weeks prior to first day of dosing on study.
* Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives or barrier methods).
* Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation.
* Symptomatic gastroparesis.
* History or evidence of use of any tobacco- or nicotine-containing product within 6 months of screening or screening quantitative urine nicotine concentration >50 ng/mL.
* Receipt of any investigational drug within 4 weeks of first day of dosing in this study.
* Any condition (intrinsic or extrinsic) that in the judgment of the Investigator will interfere with trial participation or evaluation of data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Morrow, M.D., Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States

REFERENCES:
- [Result] Hompesch M, Muchmore DB, Morrow L, Vaughn DE. Accelerated insulin pharmacokinetics and improved postprandial glycemic control in patients with type 1 diabetes after coadministration of prandial insulins with hyaluronidase. Diabetes Care. 2011 Mar;34(3):666-8. doi: 10.2337/dc10-1892. Epub 2011 Jan 27. PMID 21273493

RESULTS

PARTICIPANT FLOW:
Period: Intervention 1
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Received at Least One Dose of Study Drug | 22
Completed | 22
Not Completed | 0
Period: Washout (3 to 10 Days)
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Completed | 22
Not Completed | 0
Period: Intervention 2
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Received at Least One Dose of Study Drug | 22
Completed | 22
Not Completed | 0
Period: Washout (3 to 10 Days)
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Completed | 22
Not Completed | 0
Period: Intervention 3
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Received at Least One Dose of Study Drug | 22
Completed | 22
Not Completed | 0
Period: Washout (3 to 10 Days)
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Completed | 22
Not Completed | 0
Period: Intervention 4
Arm/Group | First Humalog+PH20, Then Humalog, Humulin-R+PH20, Humulin-R
Started | 22
Received at Least One Dose of Study Drug | 21
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of Humalog, Humulin-R, or recombinant human hyaluronidase PH20 (rHuPH20).
Groups:
- Overall Study: Humalog+recombinant human hyaluronidase PH20 (rHuPH20): Up to 3 dose-finding (DF) visits (each visit separated by 3-10 days [d]) until an appropriate dose of Humalog was identified. For each DF visit, a total of 24 units (U) of rHuPH20 was injected subcutaneously (SC) per unit of Humalog, corresponding to a mass concentration (conc) of 18.2 micrograms per milliliter (μg/mL) rHuPH20 (at final conc of 91 U/mL of Humalog)
  Humalog alone: After a 3-10 d washout (wo), a single SC injection of the appropriate identified dose of Humalog was delivered
  Humulin-R+rHuPH20: After a 3-10 d wo, up to 2 DF visits (both visits separated by 3-10 d) until an appropriate dose of Humulin-R was identified. For each DF visit, a total of 24 U of rHuPH20 was injected SC per unit of Humulin-R, corresponding to a mass conc of 20.0 μg/mL rHuPH20 (at final conc of 100 U/mL of Humulin-R)
  Humulin-R alone: After a 3-10 d wo, a single SC injection of the appropriate identified dose of Humulin-R was delivered
Arm/Group | Overall Study
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Insulin Concentration-time Curve for the First Hour (AUC0-60)
Description: AUC was derived as the area under the serum insulin concentration profile from 0 to time "t." Samples were taken 30, 20, and 10 minutes (mins) prior to treatment; every 3 mins from mins 0 through 15; and at 20, 30, 45, and 60 mins postdose.
Time Frame: Predose up to 60 minutes postdose
Population: Participants who received at least one dose of Humalog alone, Humalog + rHuPH20, Humulin-R + rHuPH20, or Humulin-R alone with evaluable AUC0-60 data.
Measure: Mean (Standard Deviation); unit: nanomole*minute per liter (nmol*min/L)
Groups:
- Humalog + rHuPH20: Humalog + recombinant human hyaluronidase PH20 (rHuPH20) was delivered for up to 3 dose-finding visits (each visit was separated by 3-10 days) until an appropriate dose of Humalog was identified. For each dose-finding visit, a total of 24 units (U) of rHuPH20 was injected subcutaneously per unit of Humalog, corresponding to a mass concentration of 18.2 micrograms per milliliter (μg/mL) rHuPH20 (at final concentration of 91 U/mL of Humalog).
- Humalog Alone: After a 3-10 day washout, a single subcutaneous injection of the appropriate identified dose of Humalog was delivered before a liquid meal.
- Humulin-R + rHuPH20: After a 3-10 day washout, Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20) was delivered for up to 2 dose-finding visits (both visits were separated by 3-10 days) until an appropriate dose of Humulin-R was identified. For each dose-finding visit, a total of 24 units (U) of rHuPH20 was injected subcutaneously per unit of Humulin-R, corresponding to a mass concentration of 20.0 micrograms per milliliter (μg/mL) rHuPH20 (at final concentration of 100 U/mL of Humulin-R).
- Humulin-R Alone: After a 3-10 day washout, a single subcutaneous injection of the appropriate identified dose of Humulin-R was delivered before a liquid meal.
Arm/Group | Humalog + rHuPH20 | Humalog Alone | Humulin-R + rHuPH20 | Humulin-R Alone
Number analyzed (Participants) | 21 | 21 | 17 | 17
nanomole*minute per liter (nmol*min/L) | 12346.67 (4996.79) [10.98 to 24.78] | 8297.62 (3670.03) | 11607.65 (6770.61) | 4331.76 (3068.10)
Statistical Analysis 1: Comparison: Humalog + rHuPH20 vs Humalog Alone; Due to the exploratory nature of this study, the sample size is not based on a formal calculation; Test type: Superiority or Other; p = 0.0011, ANOVA — Statistical testing was considered exploratory, with no adjustment for inflation of Type 1 error due to multiplicity of testing; Geometric Least Squares Means Ratio = 1.54
Statistical Analysis 2: Comparison: Humulin-R + rHuPH20 vs Humulin-R Alone; Due to the exploratory nature of this study, the sample size is not based on a formal calculation; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric Least Squares Means Ratio = 3.06

2. Secondary Outcome: Maximum Serum Insulin Concentration (Cmax)
Description: Cmax was determined as the maximum of all valid serum insulin concentration measurements for each measurement series. Samples were taken 30, 20, and 10 minutes (mins) prior to treatment; every 3 mins from mins 0 through 15; at 20, 30, and 45 mins; every 30 mins from mins 60 through 240; and every 60 minutes from mins 300 through 480 postdose.
Time Frame: Predose up to 480 minutes postdose
Population: Participants who received at least one dose of Humalog alone, Humalog + rHuPH20, Humulin-R + rHuPH20, or Humulin-R alone with evaluable Cmax data
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Humalog + rHuPH20 | Humalog Alone | Humulin-R + rHuPH20 | Humulin-R Alone
Number analyzed (Participants) | 21 | 21 | 17 | 17
Picomoles per liter (pmol/L) | 307.67 (125.73) [0.78 to 0.92] | 226.38 (85.51) | 285.88 (139.54) | 165.05 (68.98)
Statistical Analysis 1: Comparison: Humalog + rHuPH20 vs Humalog Alone; Due to the exploratory nature of this study, the sample size is not based on a formal calculation; Test type: Superiority or Other; p = 0.0057, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric Least Squares Means Ratio = 1.35
Statistical Analysis 2: Comparison: Humulin-R + rHuPH20 vs Humulin-R Alone; Due to the exploratory nature of this study, the sample size is not based on a formal calculation; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Geometric Least Squares Means Ratio = 1.66

3. Secondary Outcome: Time to Maximum Serum Insulin Concentration (Tmax)
Description: Tmax was determined as the timepoint where the maximum of all valid concentration measurements for each measurement series was observed. Samples were taken 30, 20, and 10 minutes (mins) prior to treatment; every 3 mins from mins 0 through 15; at 20, 30, and 45 mins; every 30 mins from mins 60 through 240; and every 60 minutes from mins 300 through 480 postdose.
Time Frame: Predose up to 480 minutes postdose
Population: Participants who received at least one dose of Humalog alone, Humalog + rHuPH20, Humulin-R + rHuPH20, or Humulin-R alone with evaluable tmax data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Humalog + rHuPH20 | Humalog Alone | Humulin-R + rHuPH20 | Humulin-R Alone
Number analyzed (Participants) | 21 | 21 | 17 | 17
minutes | 30.24 (8.73) | 48.57 (13.34) | 57.06 (30.83) | 116.76 (65.02)
Statistical Analysis 1: Comparison: Humalog + rHuPH20 vs Humalog Alone; Due to the exploratory nature of this study, the sample size is not based on a formal calculation; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Means Difference = -18.33
Statistical Analysis 2: Comparison: Humulin-R + rHuPH20 vs Humulin-R Alone; Due to the exploratory nature of this study, the sample size is not based on a formal calculation; Test type: Superiority or Other; p = 0.0018, ANOVA; Statistical testing was considered exploratory, with no adjustment for inflation of Type 1 error due to multiplicity of testing; Least Squares Means Difference = -62.46

4. Secondary Outcome: Area Under the Blood Glucose Time-Concentration Curve Blood Glucose (AUC[BG])
Description: AUC(BG) values are reported for participants whose blood glucose (BG) was elevated higher than 140 milligrams per deciliter (mg/dL) within 4 hours of consuming a liquid meal. Blood samples were collected at 30, 20, 10, and within 5 minutes before; at 3, 6, 9, 12, 15, 20, 25 minutes; and every 10 minutes from minute 30 to 240 postdose.
Time Frame: Predose up to 4 hours after injection of study drug
Population: Participants who received at least one dose of Humalog alone, Humalog + rHuPH20, Humulin-R + rHuPH20, or Humulin-R alone with evaluable AUC(BG) data.
Measure: Geometric Mean (90% Confidence Interval); unit: minutes*milligrams per deciliter
Arm/Group | Humalog + rHuPH20 | Humalog Alone | Humulin-R + rHuPH20 | Humulin-R Alone
Number analyzed (Participants) | 22 | 22 | 21 | 21
minutes*milligrams per deciliter | 111 [35 to 357] | 526 [164 to 1685] | 181 [57 to 581] | 1,238 [343 to 4466]

ADVERSE EVENTS:
Time Frame: Adverse event data collected from Day 1 through to the end of the study, for up to 80 days.
Arm/Group | Humalog + rHuPH20 | Humalog Alone | Humulin-R + rHuPH20 | Humulin-R Alone
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 14/22 | 15/22 | 18/22 | 18/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog + rHuPH20 (N=22) | Humalog Alone (N=22) | Humulin-R + rHuPH20 (N=22) | Humulin-R Alone (N=21)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 13 (33) | 11 (17) | 14 (39) | 14 (25)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (6) | 9 (13) | 7 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless prior written permission from the Sponsor (Halozyme) is obtained.